CLINICAL TRIAL: NCT03521531
Title: Burden and Medical Care of Sarcoma in Germany: Nationwide Cohort Study Focusing on Modifiable Determinants of Patient-Reported Outcome Measures in Sarcoma Patients
Brief Title: Burden and Medical Care of Sarcoma in Germany
Acronym: PROSa
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Markus Schuler, MD, Technische Universität Dresden
Other Study IDs: 111713
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Sarcoma
Keywords: Quality of Life; Sarcoma; Patient Reported Outcomes
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to assess the treatment situation of sarcoma patients in Germany and to investigate their potential influence on Quality of Life (and other Patient Reported Outcomes) of the affected persons. Impaired quality of life domains and factors associated with it are to be identified.

To this end, a national network of sarcoma treatment specialists and a structure for patient recruitment will be established. This care network is intended to reflect the current situation of the treatment of sarcoma patients in Germany.

ELIGIBILITY:
Inclusion Criteria:

* patients with sarcoma diagnosis according to International Classification of Diseases for Oncology (ICD-O) and World Health Organisation (WHO) classification

Exclusion Criteria:

* not mentally able to fill out questionaires
* not able to till out questionaires in German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sarcoma patients treated, diagnoses or been in aftercare in a German hospital or medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 1309 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life - EORTC QLQ-C30 | 1 year
  Measured with European Organization for Research and Treatment of Cancer Quality of Life Core Questionaire (EORTC QLQ-C30). The questionnaire consists of 30 questions assessing general quality of life issues of cancer patients. The EORTC QLQ-C30 includes 5 functional scales, measuring physical, role, emotional, cognitive, and social functioning, three multi-item symptom scales (fatigue, nausea/vomiting, and pain), and six single-item scales. High scores on the functional and global scales represent better quality of life. In contrast, high scores on the symptom scale indicate poor quality of life. Each instrument can reach values from 0-100.

SECONDARY OUTCOMES:
Pain - Intensity (BPI) | 1 year
  Measured with Brief Pain Inventory (BPI). The BPI gives two scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score consists of seven subitems rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Psychological Distress - PHQ-4 | 1 year
  Measured with the Patients Health Questionnaire (PHQ-4). The PHQ-4 comprises 4 items and consists of the diagnostic core criteria for depression (PHQ-2) and for generalized anxiety disorders (GAD-2). Each instrument can reach values from 0-6. Higher Scores are indicating higher distress.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuler, MD, Principal Investigator — Technical University Dresden, Medical Faculty; Jochen Schmitt, PhD, Principal Investigator — Technical University Dresden, Medical Faculty
Locations (1):
- University Hospital Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eichler M, Hentschel L, Singer S, Hornemann B, Hohenberger P, Kasper B, Andreou D, Pink D, Jakob J, Arndt K, Kirchberg J, Richter S, Bornhauser M, Schmitt J, Schuler MK. Distress in soft-tissue sarcoma and gastrointestinal stromal tumours patients-Results of a German multicentre observational study (PROSa). Psychooncology. 2022 Oct;31(10):1700-1710. doi: 10.1002/pon.6009. Epub 2022 Aug 18. PMID 35949152
- See also: study site with information for participating patients and about recruiting study centers (in German) — https://www.uniklinikum-dresden.de/prosastudie